CLINICAL TRIAL: NCT05848089
Title: Real-time Intervention for Suicide Risk Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Principal Investigator, Adam C. Jaroszewski, PhD, Instructor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000221
Record Dates: First submitted 2023-04-18; First posted 2023-05-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Suicidal Ideation; Suicide Attempt
Keywords: Suicide; Suicidal Ideation; Suicide Attempt
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Suicide | interventions — Cognitive Behavioral Therapy; Ecological Momentary Assessment; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) + EMA (Other): Participants will receive TAU and be prompted to complete 4x/day smartphone-based EMA surveys of negative emotion and STBs.
  Interventions: Behavioral: Ecological momentary assessment (EMA); Behavioral: Treatment as usual (TAU)
- Experimental intervention + TAU (Experimental): Participants will receive TAU plus 3 brief sessions of CBT skills, one discretionary post-discharge skills booster session, and 4x/day EMA and prompted EMI, which guides in-the-moment CBT skills practice.
  Interventions: Behavioral: Brief skills sessions plus EMI skills practice prompts; Behavioral: Ecological momentary assessment (EMA); Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Brief skills sessions plus EMI skills practice prompts — (1) Three brief treatment sessions delivering core cognitive behavioral therapy (CBT) skills (mindful emotion awareness, cognitive flexibility, and changing emotional behaviors) (during hospitalization), (2) a discretionary booster session to reinforce treatment session content (that may be offered after discharge via either phone or telehealth), and (3) ecological momentary intervention (EMI) prompts to engage in guided skills practice exercises via smartphone
  Other Names: cognitive behavioral therapy; ecological momentary intervention
  Arms: Experimental intervention + TAU
Behavioral: Ecological momentary assessment (EMA) — 4x/day brief smartphone-based EMA surveys assessing negative emotions and STBs
Behavioral: Treatment as usual (TAU) — TAU (or usual care) during hospitalization and the 28-day post-discharge period

SUMMARY:
The aim of this study is to determine whether learning three skills for managing negative emotions and receiving reminders via smartphone to practice these skills reduces how often and how intensely one experiences emotional distress and suicidal thoughts.

DETAILED DESCRIPTION:
The present study is a two-arm parallel design RCT to test the efficacy of using ecological momentary intervention (EMI) to deliver therapeutic content based on the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) - an evidence-based transdiagnostic cognitive behavioral therapy (CBT) that focuses on delivering adaptive skills for managing strong emotions. Participants in this study will be 50 adult psychiatric inpatients with recent suicidal thoughts or behaviors (STBs). Participants will be randomized to receive either the control condition, which consists of treatment as usual (TAU; n = 25) and 4x/daily daily ecological momentary assessment (EMA) of emotions and STBs, or the experimental condition, consisting of TAU, 4x/daily EMA, 3 brief sessions to deliver CBT skills (mindful emotion awareness, cognitive flexibility, and changing emotional behaviors, all drawn from the UP), one discretionary skills booster session, and EMI to prompt guided skills practice (n = 25).

Control participants will receive TAU and be prompted to complete 4x/day EMA of emotions and STBs for the duration of their hospital stay and the 28-day post-discharge period. Participants randomized to the experimental conditions will receive TAU plus three brief treatment sessions delivering core UP skills content (during inpatient stays) and a discretionary booster session to reinforce treatment sessions that may be offered after discharge via either phone or telehealth. Those in the experimental condition will also receive training to use the EMI (which prompts guided skills practice), followed by smartphone-based EMA/EMI for the duration of the inpatient stay and the 28-day post-discharge period.

ELIGIBILITY:
Inclusion Criteria:

* adult status (18+ years),
* a recent suicide attempt or any report of current suicidal ideation,
* the ability to speak and write English fluently,
* ownership of and consistent access to an internet-capable smartphone (e.g., an iPhone or Android phone), and
* providing at least one collateral contact in cases where we cannot reach the participant

Exclusion criteria:

- the presence of any factor that impairs an individual's ability to provide informed consent and comprehend and effectively participate in the study including: an inability to speak or write English fluently, the presence of gross cognitive impairment due to florid psychosis, intellectual disability, dementia, acute intoxication, or the presence of extremely agitated or violent behavior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Within-person changes in momentary self-reported intensity of suicidal urges (measured on a 11-point rating scale via ecological momentary assessment) from pre- to post-EMI | Through study completion (up to 28 days after inpatient hospital discharge)
  Overall changes in momentary self-reported intensity of suicidal urges (measured on a 11-point rating scale up to 4x/day via ecological momentary assessment) from pre- to post-EMI use, among those in the experimental condition only
Between-condition differences in momentary self-reported intensity of suicidal urges (measured on a 11-point rating scale via ecological momentary assessment) | Through study completion (up to 28 days after inpatient hospital discharge)
  Means and slopes of momentary self-reported intensity of suicidal urges (measured on a 11-point rating scale up to 4x/day via ecological momentary assessment) will be compared between the experimental and control conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Faulkner Hospital, Boston, Massachusetts, United States